CLINICAL TRIAL: NCT06634420
Title: HAELO: A Phase 3, Multinational, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of NTLA-2002 in Participants With Hereditary Angioedema (HAE)
Brief Title: HAELO: A Phase 3 Study to Evaluate NTLA-2002 in Participants With Hereditary Angioedema (HAE)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Intellia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITL-2002-CL-301
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-06

CONDITIONS: Hereditary Angioedema
Keywords: Hereditary Angioedema; NTLA-2002; HAE; HAE-C1INH-Type1 or -Type 2
MeSH Terms: conditions — Angioedemas, Hereditary

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: NTLA-2002 (Active Comparator): Arm A: NTLA-2002 (50 mg; single IV infusion)
  Interventions: Biological: NTLA-2002
- Arm B: Placebo (Placebo Comparator): Arm B: Placebo (saline; single IV infusion)
  Interventions: Biological: Normal Saline IV Administration

INTERVENTIONS:
Biological: NTLA-2002 — CRISPR/Cas9 gene editing system delivered by lipid nanoparticle (LNP) for intravenous (IV) administration
  Arms: Arm A: NTLA-2002
Biological: Normal Saline IV Administration — The administration of intravenous (IV) normal saline
  Arms: Arm B: Placebo

SUMMARY:
This Phase 3 study aims to evaluate the efficacy and safety of NTLA-2002 compared to placebo in participants with HAE.

DETAILED DESCRIPTION:
This is a multinational, multicenter, double-blind, placebo-controlled study in which approximately 60 participants will be randomized in a 2:1 ratio to receive a single IV infusion of NTLA-2002 or placebo. After the Primary Observation Period (Week 1 through Week 28), participants will have the option to receive a blinded, single IV infusion of the opposite treatment. Following the Primary Observation Period, participants will enter the Long-Term Observation Period (76 weeks), for a total of 104 weeks. Including the Screening and Run-In Period, prior to the first blinded dosing, the total study duration is approximately 28 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥16 years
2. Clinical history consistent with HAE-C1INH-Type 1 or -Type 2
3. Ability to provide evidence of HAE attacks (confirmed by the Investigator) to meet the screening requirement
4. Must agree to refrain from the use of long-term prophylactic therapies from the start of the screening period through the end of the Primary Observation Period. PI must be in agreement that it is medically acceptable for the participant to do so.
5. Must have access to, and the ability to use, on-demand medication(s) to treat potential angioedema attacks
6. Adequate chemistry and hematology measures at screening
7. Must agree not to participate in another interventional study for the duration of this trial.
8. Must be capable of providing signed informed consent. Participants 16 to < 18 years of age, whose legal guardian provides informed consent, must provide assent.
9. Must agree to follow contraception requirements

Exclusion Criteria:

1. Concurrent diagnosis of any other type of recurrent angioedema or HAE with normal C1-INH
2. Have known negative reaction or hypersensitivity to any lipid nanoparticles (LNP) component.
3. Any condition that, in the Investigator's opinion, could adversely affect the safety of the subject.
4. Unwilling to comply with study procedures.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Time-normalized number of Investigator-confirmed HAE attacks | From Week 5 through Week 28

SECONDARY OUTCOMES:
Time-normalized number of Investigator-confirmed HAE attacks requiring on-demand treatment | From Week 5 through Week 28
Time-normalized number of moderate or severe Investigator-confirmed HAE attacks | From Week 5 through Week 28
Investigator-confirmed HAE attack-free status | From Week 5 through Week 28
Change from baseline to Week 28 in AE-QoL Questionnaire total score | From baseline to Week 28
Responder status, defined as reduction from baseline of at least 50%, 70%, and 90% in time-normalized number of Investigator-confirmed HAE attacks | From Week 5 through Week 28
Time-normalized number of Investigator-confirmed HAE attacks | From Week 1 through Week 28
Time-normalized number of Investigator-confirmed HAE attacks requiring on-demand treatment | from Week 1 through Week 28
Time-normalized number of moderate or severe Investigator-confirmed HAE attacks | From Week 1 through Week 28
Investigator-confirmed HAE attack-free status | From Week 1 through Week 28
Reduction from baseline of at least 50%, 70%, and 90% in time-normalized number of Investigator-confirmed HAE attacks | From Week 1 through Week 28
Long-term prophylaxis-free status | From Week 5 through Week 104
HAE treatment-free status, defined as no usage of long-term prophylaxis or on-demand medication | From Week 5 through Week 104
Complete responder status, defined as zero Investigator-confirmed attacks with no long-term prophylaxis | From Week 5 through Week 104
Reduction in the time-normalized number of Investigator-confirmed HAE attacks after crossover treatment (Week 33 through Week 104) compared to before crossover treatment (Screening through Week 28) in participants randomized to placebo | From Week 33 through Week 104 and from Screening through Week 28

CONTACTS AND LOCATIONS:
Locations (29):
- United States (14):
  - Medical Research of Arizona, Scottsdale, Arizona
  - University of California, San Diego (UCSD), San Diego, California
  - Raffi Tachdjian MD, Inc, Santa Monica, California
  - Allergy & Asthma Clinical Research, Walnut Creek, California
  - IMMUNOe International Research Centers, Centennial, Colorado
  - Asthma & Allergy Associates, Colorado Springs, Colorado
  - University of South Florida, Tampa, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University in St. Louis, St Louis, Missouri
  - NYU Langone Health - Long Island, Mineola, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Bernstein Clinical Research Center, LLC, Cincinnati, Ohio
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - AARA Research Center, Dallas, Texas
- Australia (3):
  - Campbelltown Hospital, Campbelltown, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Canada (2):
  - University of Alberta, Edmonton, Alberta
  - Ottawa Allergy Research Corporation, Ottawa, Ontario
- France (3):
  - CHU Grenoble-Alpes - Hopital Michallon, Grenoble
  - CHU de Lille - Hopital Claude Huriez, Lille
  - AP-HM - Hopital de la Timone, Marseille
- Germany (3):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Universitaetsklinikum Frankfurt - Klinikum der Johann Wolfgang Goethe Universitaet, Frankfurt
  - Medizinische Hochschule Hannover (MHH), Hanover
- Amsterdam UMC - Locatie AMC, Amsterdam, Netherlands
- New Zealand Clinical Research (NZCR), Auckland, New Zealand
- University of Cape Town - Lung Institute - Lung Clinical Research Unit, Cape Town, South Africa
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No